CLINICAL TRIAL: NCT01194102
Title: Fit for Function: A Community Wellness Program for Persons With Stroke
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Ontario Stroke Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OSNRC-2010
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2012-10

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Physical function; Community program; Patient education; Self-management
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke Community Wellness Program (Experimental): Participants with stroke will attend a 12 week Community Wellness Program. The program consists of a Community Based Exercise Program at the YMCA (2x 1 hour exercise sessions per week with specially trained fitness instructors). They will also attend a 1 hour long "Living with Stroke" education session one time per week and an independent exercise session in the fitness centre one time per week.
  Interventions: Behavioral: Community Based Exercise Program; Other: Living with Stroke Education program; Other: YMCA membership
- Regular YMCA membership (Active Comparator): The control group will have access to YMCA facilities to use at their discretion but will not attend the Community Based Exercise Program for stroke survivors or the "Living with Stroke" education program. YMCA staff working with the control group will not receive specialized training in exercise and education for stroke survivors but will be trained on important safety precautions and contraindications to exercise after stroke.
  Interventions: Other: YMCA membership

INTERVENTIONS:
Behavioral: Community Based Exercise Program — Three supervised exercise sessions per week, including individual and group sessions aimed at strengthening, flexibility and cardiovascular exercise.
  Arms: Stroke Community Wellness Program
Other: Living with Stroke Education program — Weekly 1 hour long education sessions on living with stroke, aimed at helping participants take better care of their health after a stroke.
  Arms: Stroke Community Wellness Program
Other: YMCA membership — Participants have access to YMCA facilities along with up to 7 individual sessions with a fitness trainer.

SUMMARY:
The purpose of this study is to evaluate whether persons with stroke participating in a 12-week community based wellness program for persons who have had a stroke, experience improved mobility (6 Minute Walk Test), balance, (The Short Portable Performance Test and Timed Up and Go), strength (JAMAR hand grip dynamometry), level of physical activity (Rapid Assessment of Physical Activity), reintegration in community (Reintegration into Normal Living Index), self efficacy (Patient Activation Measure) and Quality of Life (Stroke Specific Quality of Life Scale) compared to persons who do not participate in the program.

DETAILED DESCRIPTION:
The program will be delivered through a partnership between Hamilton Health Sciences, the YMCA and McMaster University. Participants will attend the YMCA for exercise sessions several times a week and receive education on how to take care of themselves after a stroke. The staff who will deliver the program will have specialized training on how to help people with stroke to exercise safely and effectively. Control group participants will be provided with YMCA memberships but will not have access to stroke specific education and group exercise classes.

Staff assisting the control group will be trained in safety and contraindications after stroke, but will not receive the additional specialized training in exercise/education programs for persons with stroke.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18years
* living in the community
* able to ambulate ≥10 meters with or without an assistive device
* able to tolerate 60 minutes activity with rest intervals
* have clearance from a physician to participate in the program
* can independently follow instructions
* are not involved in active rehabilitation

Exclusion Criteria:

* musculoskeletal contraindications to exercise
* unstable cardiovascular conditions
* unstable medical conditions
* significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Six minute Walk Test (6MWT) | baseline, 12 weeks and 24 weeks
  The 6MWT is a test of exercise capacity that is measured as the distance walked in 6 minutes. Participants are instructed to cover as much ground as possible in 6 minutes. A greater distance walked indicates a better performance. The unit of measurement is metres.
Hand Grip Strength | baseline, 12 weeks, 24 weeks
  Hand grip strength (average of 3 trials with either hand) will be measured using a JAMAR hand-held dynamometer. Handgrip has been shown to correlate with elbow flexion strength, knee flexion strength and trunk extension strength. The unit of measurement is kilograms. Higher numbers indicate greater grip strength.
Rapid Assessment of Physical Activity (RAPA) | baseline, 12 weeks, 24 weeks
  The RAPA measures an individuals Level of Physical Activity. The RAPA is a 9 item measure that assesses frequency and intensity of aerobic physical activity and frequency of strengthening and flexibility exercises. The unit of measurement is numbers on a scale. Higher scores indicate greater levels of physical activity.

SECONDARY OUTCOMES:
Patient Activation Measure (PAM) | baseline, 12 weeks, 24 weeks
  The PAM is a 13-item measure of the patient's level of knowledge, skill and confidence for self-management of their chronic condition. The unit of measurement is numbers on a scale. Scores range from 0-100 with higher scores indicating a higher level of activation.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University
Locations (1):
- Les Chater Family YMCA, Hamilton, Ontario, Canada